CLINICAL TRIAL: NCT01051258
Title: A Study of the AeriSeal System for Lung Volume Reduction in Patients With Advanced Emphysema
Brief Title: AeriSeal System for Lung Volume Reduction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-C08-003PLVGP4-5; 03-C10-001PLV
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Emphysema; Chronic Obstructive Pulmonary Disease (COPD); Pulmonary Emphysema; Lung Diseases
Keywords: Polymeric Lung Volume Reduction (PLVR); Biologic Lung Volume Reduction (BLVR); AeriSeal; treatment; device; breathing; COPD; emphysema; heterogeneous; homogeneous; Pathologic Processes; Respiratory Tract Diseases; Lung Diseases; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema; Lung Diseases; Respiratory Aspiration; Pathologic Processes; Respiratory Tract Diseases | interventions — Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: AeriSeal System — AeriSeal System for Lung Volume Reduction
  Other Names: lung volume reduction; AeriSeal; PLVR

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AeriSeal treatment in patients with advanced emphysema.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of AeriSeal treatment in patients with advanced homogeneous and heterogeneous emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of advanced emphysema as defined by FEV1/FVC<70% predicted, FEV1 of <50% predicted, TLC > 100% predicted, and RV > 135% predicted.
* Patients must have persistent symptoms despite medical therapy and either not be candidates for Lung Volume Reduction Surgery (LVRS) or have elected not to undergo LVRS.
* Patients must be > 40 years of age, have symptoms despite medical therapy, and have none of the prespecified co-morbid conditions that could influence study outcomes or their ability to tolerate bronchoscopy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in respiratory volume/total lung capacity (RV/TLC) ratio | 12 Weeks following final treatment

SECONDARY OUTCOMES:
Change from baseline in RV/TLC ratio | 24 and 48 weeks following treatment
Change from baseline in forced expiratory volume in 1 second (FEV1) (post bronchodilator) | 12, 24, 48 weeks following treatment
Change from baseline in MRC dyspnea score | 12, 24, 48 weeks following treatment
Change from baseline in 6 minute walk test (MWT) | 12, 24, 48 weeks following treatment
Change from baseline in disease-specific health related quality of life assessment (SGRQ) | 12, 24, 48 weeks following treatment

CONTACTS AND LOCATIONS:
Locations (8):
- Otto Wagner Spital Wien Interne Lungenabteilung, Vienna, Austria
- Service de Pneumologie, Hôpital Pasteur, Centre Hospitalier Universitaire de Nice, Nice, France
- Germany (4):
  - Chefarzt Klinik für Pneumologie, Bad Berka
  - Thoraxklinik Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Medizinische Klinik und Poliklinik Klinikum Großhadern, München
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva

REFERENCES:
- [Derived] Magnussen H, Kramer MR, Kirsten AM, Marquette C, Valipour A, Stanzel F, Bonnet R, Behr J, Fruchter O, Refaely Y, Eberhardt R, Herth FJ. Effect of fissure integrity on lung volume reduction using a polymer sealant in advanced emphysema. Thorax. 2012 Apr;67(4):302-8. doi: 10.1136/thoraxjnl-2011-201038. Epub 2012 Feb 28. PMID 22374920
- See also: Related Info — http://www.aerist.com